CLINICAL TRIAL: NCT04033406
Title: A Phase 1, Randomized, Placebo-Controlled Study to Evaluate the Safety, Pharmacokinetics, and Immunogenicity of VIR-2482 for the Prevention of Influenza A Illness
Brief Title: Study of VIR-2482 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vir Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VIR-2482-3001
Record Dates: First submitted 2019-07-22; First posted 2019-07-26 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Influenza A
Keywords: Influenza A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VIR-2482 (Experimental): VIR-2482
  Interventions: Drug: VIR-2482
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VIR-2482 — VIR-2482 given by intramuscular injection
  Arms: VIR-2482
Drug: Placebo — Sterile normal saline (0.9% NaCl) given by intramuscular injection
  Arms: Placebo

SUMMARY:
This is a phase 1 study in which healthy volunteers will receive VIR-2482 or placebo and will be assessed for safety, pharmacokinetics, and immunogenicity of VIR-2482 in preventing Influenza A illness.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Male or Female age 18 to < 65 years
* Body mass index (BMI) of 18.0 kg/m^2 to 32.0kg/m^2

Exclusion Criteria:

* Any clinically significant chronic or acute medical condition that makes the volunteer unsuitable for participation
* History of influenza-like illness or confirmed influenza infection within 3 months prior to randomization.
* Fever-like illness within 5 days of randomization.
* History or clinical evidence of conditions considered high risk for developing influenza-related complications.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events. | Up to 12 months post-dose
Number of participants with abnormalities in vital signs. | Up to 12 months post-dose
Number of participants with abnormalities in electrocardiogram (ECG). | Up to 12 months post-dose
Number of participants with abnormalities in clinically significant laboratory findings. | Up to 12 months post-dose

SECONDARY OUTCOMES:
Concentrations of VIR-2482 in serum | Up to 12 months post-dose
Incidence of anti-drug antibody (ADA) to VIR-2482 | Up to 12 months post-dose
Titers (if applicable) of anti-drug antibody (ADA) to VIR-2482 | Up to 12 months post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- Investigative Site, Brisbane, Queensland, Australia

REFERENCES:
- [Derived] Plotnik D, Sager JE, Aryal M, Fanget MC, Peter A, Schmid MA, Cebrik D, Mogalian E, Boundy K, Yeh WW, Griffin P, Reyes M. A phase 1 study in healthy volunteers to investigate the safety, tolerability, and pharmacokinetics of VIR-2482: a monoclonal antibody for the prevention of severe influenza A illness. Antimicrob Agents Chemother. 2024 Apr 3;68(4):e0127323. doi: 10.1128/aac.01273-23. Epub 2024 Feb 20. PMID 38376227